CLINICAL TRIAL: NCT06783426
Title: Older Adults' Experiences of Oral Rehabilitation - a Qualitative Interview Study
Status: Completed | Type: Observational
Sponsor: Folktandvården Stockholms län AB (Other Government)
Responsible Party: Sponsor
Other Study IDs: FTV 2407-0291
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Oral Health
Keywords: Qualitative study; Interview study; Quality of Life; Patient experience; oral rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults who have undergone extensive oral rehabilitation: The cohort includes older adults, who have been referred to the Eastman Institute in Stockholm for extensive oral prosthetic rehabilitation. They have previously agreed to participate in the intervention study "Cognitive changes and neural correlates after oral rehabilitation procedures in older adults" at the Eastman Institute in Stockholm . The oral rehabilitation usually includes fixed prosthodontics. These patients are asked to participate in one interview after their treatment is completed to share their experiences before, during, and after the treatment.

SUMMARY:
The aim of this study is to gain knowledge and understanding about older adults' experiences of comprehensive oral prosthetic rehabilitation and their life situation before, during and after the treatment. This is both to deepen the knowledge gained in an ongoing interventional study, but also to increase the understanding of how to best meet older adults' needs when planning and performing oral rehabilitation in any dental surgery.

DETAILED DESCRIPTION:
This qualitative study will be based on individual, semi-structured interviews using an Interview Guide focusing on the participants´ perceptions, experiences, and reflections. The interviews will then be analyzed with a descriptive content analysis method according to Graneheim and Lundman.

ELIGIBILITY:
Inclusion Criteria:

* Completed prosthetic treatment in the original study 2-12 months ago
* Age 65-80 years at start of the original study
* Masticatory dysfunction (Eichner's index B3-B4 or C1-C4) for original study
* Mini-Mental-State-Examination-test (MMSE) score >26 for original study

Exclusion criteria for the original study:

* Neuropsychological disease
* Severely impaired hearing or vision
* Poor knowledge of the Swedish language
* Having had a stroke ≤ 6 months before inclusion

No additional exclusion criteria for our study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The participants have been assessed with comprehensive quantitative methods of their neuropsychological status, oral function, and quality of life in conjunction with the original study from which they were recruited. They were then treated with oral prosthetic therapy and are reassessed at a follow-up three months after completion of the therapy. Our participants are recruited consecutively as they finish treatment at the Eastman Institute until we consider to have obtained "saturation" of our results.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
The participants perceived experiences | 3-9 months after completing the prosthetic treatment.
  Since this is a qualitative study, we have no traditional outcome measures. Instead, completing the interview and sharing their perceived experiences during the treatment procedure , how their oral health may have affected their life situation, their quality of life and well-being before, during and after the treatment may serve as our primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotta Elleby, PhD, DDS, Principal Investigator — Folktandvården Stockholm
Locations (1):
- Folktandvården Stockholms Län AB, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Our recordings of the interviews may contain sensitive data, and the participants could be identified by voice. According to the approved ethical application we are not supposed to share any data that can be used to identify the participants. However, it is possible that the de-identified transcriptions of the interviews could be shared.

REFERENCES:
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Elgestad Stjernfeldt P, Faxen-Irving G, Wardh I. Masticatory ability in older individuals: A qualitative interview study. Gerodontology. 2021 Jun;38(2):199-208. doi: 10.1111/ger.12515. Epub 2020 Nov 27. PMID 33245159
- [Background] Hyland R, Ellis J, Thomason M, El-Feky A, Moynihan P. A qualitative study on patient perspectives of how conventional and implant-supported dentures affect eating. J Dent. 2009 Sep;37(9):718-23. doi: 10.1016/j.jdent.2009.05.028. Epub 2009 Jun 7. PMID 19559515
- [Background] Trulsson U, Engstrand P, Berggren U, Nannmark U, Branemark PI. Edentulousness and oral rehabilitation: experiences from the patients' perspective. Eur J Oral Sci. 2002 Dec;110(6):417-24. doi: 10.1034/j.1600-0722.2002.21394.x. PMID 12507214
- [Background] Nordenram G, Davidson T, Gynther G, Helgesson G, Hultin M, Jemt T, Lekholm U, Nilner K, Norlund A, Rohlin M, Sunnegardh-Gronberg K, Tranaeus S. Qualitative studies of patients' perceptions of loss of teeth, the edentulous state and prosthetic rehabilitation: a systematic review with meta-synthesis. Acta Odontol Scand. 2013 May-Jul;71(3-4):937-51. doi: 10.3109/00016357.2012.734421. Epub 2012 Oct 29. PMID 23101439
- [Background] Hedberg L, Ekman U, Nordin LE, Smedberg JI, Skott P, Seiger A, Sandborgh-Englund G, Westman E, Kumar A, Trulsson M. Cognitive changes and neural correlates after oral rehabilitation procedures in older adults: a protocol for an interventional study. BMC Oral Health. 2021 Jun 9;21(1):297. doi: 10.1186/s12903-021-01654-5. PMID 34107933